CLINICAL TRIAL: NCT03828500
Title: Preoperative Fasting for Ambulatory Cataract Surgery: A Time-Interrupted Prospective Study
Brief Title: Preoperative Fasting for Ambulatory Cataract Surgery: The PRACTICE Study
Acronym: PRACTICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Sherif El-Defrawy, Chair and Professor of Department of Ophthalmology and Vision Sciences, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRACTICE_2019_001
Record Dates: First submitted 2019-01-30; First posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Cataract Extraction; Fasting; Aspiration Pneumonitis
Keywords: Cataract; Cataract Extraction; Fasting; Preoperative Period; Interrupted Time Series Analysis; Guideline; Patient Care
MeSH Terms: conditions — Fasting; Pneumonia, Aspiration; Cataract

STUDY DESIGN:
Masking Description: Not masked
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Arm (Experimental): encouraged by Research Assistant to drink clear fluids up to 2 hour limit. Arm 2 - standard of care
  Interventions: Behavioral: Assistant-encouraged fasting up to ASA/CAS guideline limits
- Control Arm (No Intervention)

INTERVENTIONS:
Behavioral: Assistant-encouraged fasting up to ASA/CAS guideline limits — Research Assistant encourages patient to drink clear fluids up to 2 hour limit before surgery, in accordance with the latest ASA and CAS guidelines.
  Arms: Experimental Arm

SUMMARY:
The current standard for cataract surgery is phacoemulsification with intraocular lens (IOL) implantation. In this procedure, topical anesthesia has become favoured over local anesthetic blocks due to potential serious complications resulting from retrobulbar or peribulbar anesthesia. Routinely, intravenous sedation is used to supplement the topical anesthesia. If patients are not fasted, there is the potential to reduce preoperative discomfort and anxiety, ultimately improving the satisfaction with the care received. An additional benefit is that liberal fasting policies allow for flexibility in the scheduling of cases, particularly for urgent or semi-urgent situations. Clinical practice guidelines for cataract surgery published by the Canadian Ophthalmological Society (COS) recommend that fasting is unnecessary if only topical anesthesia is used without intravenous (IV) opiates or sedation. In general, these suggestions are in agreement with guidelines from the United Kingdom's Royal College of Ophthalmologists, who note that "it is unnecessary to fast patients for local anesthetic cataract surgery." According to the CAS practice guidelines, the same fasting restrictions are applied when IV sedation or anesthesia with peripheral nerve blocks (e.g. retrobulbar or peribulbar blocks) are administered. At our centre at the Kensington Eye Institute (KEI) in Toronto, Canada, almost all cataract patients receive fentanyl and midazolam, with propofol given only in rare circumstances with close observation.

This research project at the Kensington Eye Institute will consist of two phases, namely a prospective, consecutive observational analysis and a prospective time-interrupted study. In the first phase, an observational analysis will be conducted in which consecutive cataract surgery patients will be surveyed with a validated questionnaire to assess their satisfaction. Inclusion criteria will include any cataract patient scheduled for surgery who is willing and able to participate in the study, with fully informed consent provided.

Previously published literature has evaluated the use of a patient satisfaction questionnaire regarding preoperative fasting, which includes items on hunger, thirst, hoarseness of voice, difficulty breathing, pain, agitation, anxiety, nausea, vomiting, shivering and problems with concentration. A Research Assistant will complete the questionnaire with all patients preoperatively at KEI, as well as a baseline demographic checklist that will include the patient's age, gender, laterality, surgeon, length of time fasted for solids and clear liquids, as well as the type and amount of solids and liquids. Secondary endpoints will be collected postoperatively and will include the incidence of aspiration, nausea and vomiting, as well as the rate of cancellations of surgeries directly related to issues with fasting guidelines. The first phase of the study will be used to conduct an appropriate sample size calculation, which will ensure that our second phase is not underpowered for the primary efficacy endpoint.

In the second phase, a time-interrupted prospective study will be established with the following two arms: (1) experimental arm: patients will be encouraged by the Research Assistant to drink clear fluids right up to the 2 hour limit as specified in the latest ASA and CAS guidelines, with no intervention applied for solids, and (2): control arm: standard of care without any encouragement to drink clear fluids up to the 2 hour limit. Patients will be assigned to groups based on month, so that the first month of study execution will enroll all patients into the experimental arm, the second month will enroll only into the control arm, and that subsequent months will alternate enrollment in a similar method.

Given the design, the study will be in accordance with the latest ASA and CAS preoperative fasting guidelines, and will not involve any use of financial or other methods of coercion to incentivize patients that are randomly assigned to the experimental arm. The encouragement process will only involve the Research Assistant asking and encouraging the patient to drink a standardized quantity of clear fluid (up to 400mL of water, coffee, tea, apple or cranberry juice and maximum of 2 teaspoons of sugar) up to the ASA and CAS mandated guideline of 2 hours preoperatively, with the patient making the final determination of whether to comply. Following the encouragement process, a demographics and satisfaction questionnaire will be administered to each patient preoperatively, as well as another satisfaction questionnaire administered following the surgery. Baseline demographics, primary and secondary endpoints will remain consistent with the first phase.

ELIGIBILITY:
Inclusion Criteria:

* any cataract patient scheduled for surgery at the Kensington Eye Institute who is willing and able to participate in the study, with fully informed consent provided.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-01-31 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Demographic baseline parameters | Immediately post-operatively
  Patient number, age, gender, surgery on left or right eye, surgeon, fasting time - solids (hours), fasting time - clear liquids (hours), solid foods eaten in last 24 hours, liquids drank in last 24 hours
Satisfaction Questionnaire | Immediately post-operatively
  Hunger, thirst, voice hoarseness, difficulty breathing, pain, agitation, anxiety, nausea, vomiting, shivering, difficulty in concentration
  Scale name: patient satisfaction with preoperative fasting questionnaire
  For this scale, the following choices will be provided for each item: strongly agree, agree, neutral, disagree, strongly disagree.
  Strongly agree and agree options represent a worse outcome. Strongly disagree and disagree options represent a better outcome.
  The scores from individual items will be averaged to yield a total score.

SECONDARY OUTCOMES:
Regarding patient satisfaction survey | Immediately post-operatively
  The proportion of participants that believe the survey is effective, clear, relevant, simple and consistent in measuring distress and burden of preoperative fasting. The number of participants that suggest further questions to add to the existing survey.

OTHER OUTCOMES:
Rates of postoperative aspiration | Immediately post-operatively
  The proportion of patients in sample sustaining aspiration postoperatively.
Rates of cancellation of surgery due to preoperative fasting requirement violation | Immediately post-operatively
  The proportion of cataract surgery patients at the surgical centre in the study timeframe needing to have surgery cancelled due to preoperative fasting requirement violation

CONTACTS AND LOCATIONS:
Overall Officials: Sherif El-Defrawy, MD, PhD, FRCSC, Principal Investigator — Kensington Eye Institute
Locations (1):
- Kensington Eye Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hosoda Y, Kuriyama S, Jingami Y, Hattori H, Hayashi H, Matsumoto M. A comparison of patient pain and visual outcome using topical anesthesia versus regional anesthesia during cataract surgery. Clin Ophthalmol. 2016 Jun 20;10:1139-44. doi: 10.2147/OPTH.S109360. eCollection 2016. PMID 27382247
- [Background] Smith R. Cataract extraction without retrobulbar anaesthetic injection. Br J Ophthalmol. 1990 Apr;74(4):205-7. doi: 10.1136/bjo.74.4.205. PMID 2337544
- [Background] Pandey SK, Werner L, Apple DJ, Agarwal A, Agarwal A, Agarwal S. No-anesthesia clear corneal phacoemulsification versus topical and topical plus intracameral anesthesia. Randomized clinical trial. J Cataract Refract Surg. 2001 Oct;27(10):1643-50. doi: 10.1016/s0886-3350(01)00793-3. PMID 11687365
- [Background] Canadian Ophthalmological Society Cataract Surgery Clinical Practice Guideline Expert Committee. Canadian Ophthalmological Society evidence-based clinical practice guidelines for cataract surgery in the adult eye. Can J Ophthalmol. 2008 Oct;43 Suppl 1:S7-57. doi: 10.1139/i08-133. No abstract available. English, French. PMID 19177161
- [Background] Royal College of Ophthalmologists. Cataract Surgery Guidelines. London, UK: Royal College of Ophthalmologists, 2004.
- [Background] Dobson G, Chong M, Chow L, Flexman A, Kurrek M, Laflamme C, Lagace A, Stacey S, Thiessen B. Guidelines to the Practice of Anesthesia - Revised Edition 2018. Can J Anaesth. 2018 Jan;65(1):76-104. doi: 10.1007/s12630-017-0995-9. Epub 2017 Dec 14. PMID 29243160
- [Background] Bopp C, Hofer S, Klein A, Weigand MA, Martin E, Gust R. A liberal preoperative fasting regimen improves patient comfort and satisfaction with anesthesia care in day-stay minor surgery. Minerva Anestesiol. 2011 Jul;77(7):680-6. Epub 2009 Feb 4. PMID 19190563
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707